CLINICAL TRIAL: NCT05975749
Title: A Study of Compared Adjuvant Serplulimab and Trastuzuma and Chemotherapy vs Chemotherapy Only in Her-2 Positive Gastric Cancer With II-III Stage Following Curative Resection
Brief Title: Adjuvant Serplulimab and Trastuzuma and Chemotherapy in Her-2+ Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-her2
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Adjuvant treatment; Trastuzuma; Serplulimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Treatment of Serplulimab and Trastuzuma and Chemotherapy (Experimental)
  Interventions: Drug: Serplulimab; Drug: Trastuzuma; Drug: Chemotherapy
- Adjuvant Chemotherapy only (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Serplulimab — Serplulimab: 4.5mg/Kg on day 1
  Arms: Adjuvant Treatment of Serplulimab and Trastuzuma and Chemotherapy
Drug: Trastuzuma — Trastuzuma: 8mg/Kg ( the first cycle)，6mg/Kg (the rest of cycles) on day 1
  Arms: Adjuvant Treatment of Serplulimab and Trastuzuma and Chemotherapy
Drug: Chemotherapy — Chemotherapy: Capecitabine or S-1 and Oxaliplatin (eight 3-week cycles of oral capecitabine 1000 mg/m² or S-1 40 mg/m2 twice daily on days 1-14 plus intravenous oxaliplatin 130 mg/m² on day 1) for 6 months or progress of disease

SUMMARY:
The purpose of this study is to find out whether treatment with Serplulimab combined with Trastuzumab and Chemotherapy will improve the survival of gastric cancer patients with stage II-III after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 20 years old and upper age limit of 80 years old.
2. Be proven to be primary adenocarcinoma of gastric cancer and staged II-III by pathological evidences
3. R0 gastrectomy with D2 lymphadenectomy
4. Her2+ diagnosed by Immunohistochemistry or FISH
5. ECOG (ECOG score standard) performance status of 0 or 1 and expected to survive more than 6 months
6. No contraindications, including normal peripheral blood routine, liver and kidney function and electrocardiogram （WBC≥3.5 x 109 /L, NEU≥1.2 x 109 /L,PLT≥90 x 109 /L and HGB≥80g/L).

Exclusion Criteria:

1. Patients with stage I and IV.
2. Unavailable for R0 resection and D2 lymph node dissection.
3. Multiple primary tumors
4. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases.
5. History of chemotherapy, radiotherapy, immunotherapy or target therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year
  DFS

SECONDARY OUTCOMES:
Overall survival | 3-year
  OS
Side effects | 12 months]
  Complications such as Nausea, vomiting, myelosuppression and Liver or kidney function disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No